CLINICAL TRIAL: NCT02211365
Title: Registro Campania Salute Network for the Treatment of Hypertension and Correlated Diseases
Brief Title: Registro Campania Salute Network on Hypertension
Acronym: RCSN
Status: Recruiting | Type: Observational
Sponsor: Federico II University (Other)
Responsible Party: Principal Investigator, RAFFAELE IZZO, Professor, Federico II University
Other Study IDs: 16/14
Record Dates: First submitted 2014-04-08; First posted 2014-08-07 (Estimated); Last update posted 2025-08-08 (Actual); Status verified 2025-08

CONDITIONS: Hypertension; Heart Disease, Hypertensive
Keywords: Hypertension; CVD
MeSH Terms: conditions — Hypertension; Heart Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The Registro Campania Salute Network (RCSN) is a prospective registry aimed at improving the management of essential hypertension by integrating the activity of general practitioners (GPs) with that of the hypertension specialist. It involves selected GPs homogeneously allocated in the regional area, and the Hypertension Clinic of the Federico II University in Naples, which served as co-ordinating centre. Through the RCSN system it is possible to store clinical data detected at each visit between the peripheral units and the co-ordinating centre and to support scientific analysis of the dataset.

DETAILED DESCRIPTION:
The patients will be followed over a period of twenty years and all clinical data will be recorded in order to investigate the role of hypertension and correlated disease on this patient population

ELIGIBILITY:
Inclusion Criteria:

-Hypertension

* 18 years old

Exclusion Criteria:

* Refused to sign informed consent

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hypertensive patients
Sampling Method: Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2014-02 (Actual); Primary Completion 2017-03 (Actual); Study Completion 2030-04 (Estimated)

PRIMARY OUTCOMES:
MACCE | every year up to 20 years
  Major adverse cardiac and cerebrovascular events

CONTACTS AND LOCATIONS:
Overall Officials: Bruno Trimarco, MD, Principal Investigator — Dipartimento di Scienze Biomediche Avanzate, Università degli Studi di Napoli Federico II
Locations (1):
- Department od advanced biomedical sciences, Università degli studi di Napoli Federico II, Via sergio Pansini 5, Napoli, Napoli, Italy

REFERENCES:
- [Derived] Mancusi C, Basile C, Gerdts E, Fucile I, Manzi MV, Lembo M, Pacella D, Giugliano G, Canciello G, Piccolo R, Spinelli A, Morisco C, De Luca N, Trimarco B, de Simone G, Bossone E, Izzo R, Losi MA, Esposito G. Carotid plaque offsets sex-related differences in cardiovascular risk of young hypertensive patients. Eur J Intern Med. 2024 Dec;130:137-143. doi: 10.1016/j.ejim.2024.09.007. Epub 2024 Sep 17. PMID 39294033
- [Derived] Trimarco V, Manzi MV, Izzo R, Mone P, Lembo M, Pacella D, Esposito G, Falco A, Morisco C, Gallo P, Santulli G, Trimarco B. The therapeutic concordance approach reduces adverse drug reactions in patients with resistant hypertension. Front Cardiovasc Med. 2023 May 5;10:1137706. doi: 10.3389/fcvm.2023.1137706. eCollection 2023. PMID 37215551
- [Derived] Lembo M, Acampa W, Rao MAE, Manzi MV, Morisco C, Esposito G, Assante R, Zampella E, Nappi C, Gaudieri V, Mannarino T, Mancusi C, de Simone G, Izzo R, Cuocolo A, Trimarco B. Left Ventricular Mechano-Energetic Efficiency Identifies an Early Impairment of Myocardial Blood Flow in Arterial Hypertension. Hypertension. 2023 Jul;80(7):1534-1543. doi: 10.1161/HYPERTENSIONAHA.123.21071. Epub 2023 May 12. PMID 37170833
- [Derived] Stabile E, Franzese M, Chianese S, Alfani A, Gerardi D, Colaiori I, Annunziata M, Nappi P, Scalise M, Di Serafino L, Puzone B, Avvedimento M, Leone A, Ilardi F, Piccolo R, Franzone A, Cirillo P, Morisco C, Trimarco B, Esposito G. Predictors of adherence to composite therapy after acute coronary syndromes. J Cardiovasc Med (Hagerstown). 2021 Aug 1;22(8):645-651. doi: 10.2459/JCM.0000000000001201. PMID 33966020
- [Derived] Mancusi C, Losi MA, Albano G, De Stefano G, Morisco C, Barbato E, Trimarco B, De Luca N, de Simone G, Izzo R. Characteristics and Outcomes of Patients Presenting With Hypertensive Urgency in the Office Setting: The Campania Salute Network. Am J Hypertens. 2020 Apr 29;33(5):414-421. doi: 10.1093/ajh/hpaa003. PMID 31930302
- [Derived] Canciello G, Mancusi C, Losi MA, Izzo R, Trimarco B, de Simone G, De Luca N. Aortic Root Dilatation Is Associated With Incident Cardiovascular Events in a Population of Treated Hypertensive Patients: The Campania Salute Network. Am J Hypertens. 2018 Nov 13;31(12):1317-1323. doi: 10.1093/ajh/hpy113. PMID 30099532
- [Derived] Mancusi C, Izzo R, Ferrara LA, Rozza F, Losi MA, Canciello G, Pepe M, de Luca N, Trimarco B, de Simone G. Is increased uric acid a risk factor or a defensive response? The Campania Salute Network. Nutr Metab Cardiovasc Dis. 2018 Aug;28(8):839-846. doi: 10.1016/j.numecd.2018.04.013. Epub 2018 May 4. PMID 29898822
- [Derived] Izzo R, Losi MA, Stabile E, Lonnebakken MT, Canciello G, Esposito G, Barbato E, De Luca N, Trimarco B, de Simone G. Development of Left Ventricular Hypertrophy in Treated Hypertensive Outpatients: The Campania Salute Network. Hypertension. 2017 Jan;69(1):136-142. doi: 10.1161/HYPERTENSIONAHA.116.08158. Epub 2016 Nov 28. PMID 27895192